CLINICAL TRIAL: NCT05383781
Title: Effect of Adding Short Foot Exercise to Hip and Knee Focused Exercises in Treatment of Patients With Patellofemoral Pain Syndrome
Brief Title: Effect of Short Foot Exercise in Treatment of Patients With Patellofemoral Pain Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Abdallah Mohamed Kamel Mohamed Ali, Principal Investigator -Assistant lecturer at Faculty of Physical Therapy, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P.T.REC/012/003641
Record Dates: First submitted 2022-05-13; First posted 2022-05-20 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: Short foot exercise; Patellofemoral pain syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Papaverine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hip and Knee exercise group (Active Comparator): Individuals in this group will perform exercises for the Hip and knee only.
  Interventions: Other: Hip and Knee focused exercises
- Hip , Knee exercise and SFE group (Experimental): Individuals in this group will perform exercises for Hip , knee and also short foot exercise
  Interventions: Other: Hip and Knee focused exercises; Other: Short foot exercise

INTERVENTIONS:
Other: Hip and Knee focused exercises — Exercises which improves muscle strength, ROM
Other: Short foot exercise — The 'short foot exercise' has been described as a means to isolate contraction of the plantar intrinsic muscles.
  Arms: Hip , Knee exercise and SFE group

SUMMARY:
Purposes of the study

To investigate the effect of adding Short foot exercise on patellofemoral pain syndrome on knee Pain, Function, Balance and abductors, quadriceps Muscle strength.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as PFPS
* Pain elicited at least by two of the following four tests; (i) Isometric muscle contraction with slight bent knee,(ii) palpation of the patellofemoral joint line, (iii) patellar compression against the femoral bone (iv) active resisted knee extension.
* Psychological and mentally stable
* No previous knee surgery, except for diagnostic arthroscopy.
* No current knee pathologies (e.g. osteoarthritis)
* Navicular drop test more than 10 mm which indicated pronated foot

Exclusion Criteria:

- Subjects will be excluded if they don't meet the inclusion criteria.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
assessment of knee pain | Change from baseline pain at 6th week
  by visual analogue scale ( VAS ) to assess knee pain -minimum score is 0 point and maximum score is 10. score of 10 means worst pain outcome
assessment of knee function | Change from baseline function at 6th week
  by Anterior Knee Pain Scale ( AKP )- minimum score is 0 point and maximum score is 100 points . score of 100 means no pain . this scale assesses knee pain and function

SECONDARY OUTCOMES:
Assessment of muscle strength | Change from baseline at 6th week
  by Hand-Held Dynamometer (HHD):
Assessment of balance: | Change from baseline at 6th week
  by Biodex Balance System is the device to assess balance and postural stability .

CONTACTS AND LOCATIONS:
Overall Officials: Abdallah Ali, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kamel AM, Ghuiba K, Abd Allah DS, Fayaz NA, Abdelkader NA. Effect of adding short foot exercise to hip and knee focused exercises in treatment of patients with patellofemoral pain syndrome: a randomized controlled trial. J Orthop Surg Res. 2024 Apr 1;19(1):207. doi: 10.1186/s13018-024-04688-x. PMID 38561773